CLINICAL TRIAL: NCT02610127
Title: Post-Marketing Non-Interventional Safety Evaluation of Obizur in the Treatment of Bleeding Episodes for Patients With Acquired Hemophilia A
Status: Completed | Type: Observational
Sponsor: Baxalta now part of Shire (Industry)
Collaborators: Baxalta Innovations GmbH, now part of Shire (Industry)
Responsible Party: Sponsor
Organization: Takeda (Industry)
Other Study IDs: 241302; EUPAS36659 (Registry Identifier: EUPAS)
Record Dates: First submitted 2015-10-29; First posted 2015-11-20 (Estimated); Last update posted 2021-08-05 (Actual); Status verified 2021-08

CONDITIONS: Acquired Hemophilia A
MeSH Terms: conditions — Factor 8 deficiency, acquired | interventions — Factor VIII

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- OBIZUR - Prospective Participants: Participants enrolled and treated with Obizur after the prospective study start date
  Interventions: Biological: OBIZUR
- OBIZUR - Retrospective Participants: Retrospective chart review of participants treated with OBIZUR from product approval date until prior to the prospective study start date
  Interventions: Biological: OBIZUR

INTERVENTIONS:
Biological: OBIZUR — Treating physician will determine treatment regimen, frequency of laboratory and clinical assessments, according to routine clinical practice.
  Other Names: rpFVIII; Recombinant pFVIII; Antihemophilic Factor (Recombinant); Porcine Sequence

SUMMARY:
The overall objective is to enroll patients with acquired hemophilia A (AHA) who are prescribed and treated with Obizur, to assess safety, and to describe factors related to safety, utilization and effectiveness in a real-world setting.

DETAILED DESCRIPTION:
This study is a multi-center, uncontrolled, open-label, non-interventional post-marketing safety surveillance study to describe the use of Obizur in patients with acquired hemophilia A (AHA), and secondarily, where data are available, to describe the hemostatic effectiveness and immunogenicity of Obizur.

Patients should be enrolled at the earliest possible time point after initiating Obizur.

In an attempt to collect safety and utilization data on patients treated with Obizur since Food and Drug Administration (FDA) approval in October 2014, Baxalta will make an effort to identify all persons treated with Obizur and to collect data for as many patients as possible.

ELIGIBILITY:
Inclusion Criteria:

1. Participant is ≥18 years of age at the time of informed consent.
2. Participant has AHA, and is being treated/was treated with Obizur.
3. Participant or the participant's legally authorized representative is willing and able to provide informed consent, unless informed consent is not required

Exclusion Criteria:

1. Participant has a known anaphylactic reaction to the active substance, to any of the excipients, or to hamster protein.
2. Participant has a concomitant bleeding disorder(s) other than acquired hemophilia A (AHA).
3. Participant has participated in another clinical study involving a medicinal product or device within 30 days prior to enrollment or is scheduled to participate in another clinical study involving a medicinal product or device during the course of the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 53 (Actual)
Dates: Start 2015-12-30 (Actual); Primary Completion 2019-06-07 (Actual); Study Completion 2019-06-07 (Actual)

PRIMARY OUTCOMES:
Incidence of therapy-related SAEs and level of severity | Throughout the study period of approximately 4 years

SECONDARY OUTCOMES:
Hemostatic effectiveness assessment for resolution of bleeding | Throughout the study period, up to approximately 4 years
  Determined as either bleeding stopped or did not stop
Time to bleeding resolution, participant study termination, or switch to another treatment | Throughout the study period, up to approximately 4 years
Number of Obizur units/kg required for control of bleeding | Throughout the study period, up to approximately 4 years
Number of Obizur infusions required for control of bleeding | Throughout the study period, up to approximately 4 years
Titer of newly recognized anti-porcine Factor VIII (anti-pFVIII) neutralizing antibodies (inhibitors) or increase in titer of anti-pFVIII inhibitors from baseline and changes over time. | Throughout the study period of approximately 4 years
Impact of the inhibitor on hemostatic efficacy and any associated clinical manifestations. | Throughout the study period of approximately 4 years
Occurrence of hypersensitivity reactions | Throughout the study period of approximately 4 years
Occurrence of any thrombogenic event | Throughout the study period of approximately 4 years

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, Study Director — Shire
Locations (16):
- United States (16):
  - University of Colorado Health, Aurora, Colorado
  - University of Florida, Gainesville, Florida
  - Emory University School of Medicine, Atlanta, Georgia
  - Bleeding and Clotting Disorders Institute, Peoria, Illinois
  - Indiana Hemophilia and Thrombosis Center, Indianapolis, Indiana
  - University of Iowa Hospitals & Clinics, Iowa City, Iowa
  - Tulane University Hospital & Clinics, New Orleans, Louisiana
  - Henry Ford Health System, Detroit, Michigan
  - Michigan State University, East Lansing, Michigan
  - Washington University, St Louis, Missouri
  - Duke University Medical Center, Durham, North Carolina
  - Comprehensive Cancer Center of Wake Forest Unversity, Winston-Salem, North Carolina
  - Cleveland Clinic, Cleveland, Ohio
  - University of Pennsylvania Health System, Philadelphia, Pennsylvania
  - University of Utah Health Sciences Center, Salt Lake City, Utah
  - Blood Center of Southeast Wisconsin, Milwaukee, Wisconsin

IPD SHARING:
Plan to Share IPD: Yes
Takeda provides access to the de-identified individual participant data (IPD) for eligible studies to aid qualified researchers in addressing legitimate scientific objectives (Takeda's data sharing commitment is available on https://clinicaltrials.takeda.com/takedas-commitment?commitment=5). These IPDs will be provided in a secure research environment following approval of a data sharing request, and under the terms of a data sharing agreement.
Supporting Information: Study Protocol, SAP, ICF, CSR
Access Criteria: IPD from eligible studies will be shared with qualified researchers according to the criteria and process described on https://vivli.org/ourmember/takeda/. For approved requests, the researchers will be provided access to anonymized data (to respect patient privacy in line with applicable laws and regulations) and with information necessary to address the research objectives under the terms of a data sharing agreement.
URL: https://vivli.org/ourmember/takeda/

REFERENCES:
- See also: To obtain more information on the study, click here/on this link — https://clinicaltrials.takeda.com/study-detail/5f6b5fc64db2bf003ab45d33